CLINICAL TRIAL: NCT02124005
Title: Evaluation of the Minimum Effective Concentration of Bupivacaine (EC50) in Femoral Block for Analgesia by Ultrasound After Knee Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ed Carlos Rey Moura (Other)
Responsible Party: Sponsor-Investigator, Ed Carlos Rey Moura, doctor, Federal University of São Paulo
Organization: Federal University of São Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EC50 femoral block bupivacaine
Record Dates: First submitted 2014-04-13; First posted 2014-04-28 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Knee Surgery; Postoperative Pain
Keywords: Knee surgery; Femoral block; Bupivacaine; Ultrasound
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Femoral block, ultrasound, bupivacaine (Experimental)
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine

SUMMARY:
The purpose of the study is to determine the minimum effective concentration of bupivacaine (EC50) in femoral block for analgesia by ultrasound after knee surgery.

DETAILED DESCRIPTION:
45 patients classified as ASA P1 or P2 aged between 18 and 65 candidates for elective knee operation via arthroscopy were included in the study. All patients received femoral nerve block guided by ultrasound with bupivacaine, 22 ml. The first patient at a concentration of 0.25%. The other patients with higher or lower concentrations if the first patient has pain> 3 or <3 on visual analogic scale respectively after awakening of surgical anesthesia. For surgical anesthesia each patient will undergo general anesthesia. At the end of the surgical procedure and anesthetic awakening patients will be evaluated for analgesia by verbal numeric scale. The modified Dixon method was used to find the EC50 and EC95 of bupivacaine for analgesia of femoral nerve block guided by ultrasound. Concentration still correlated with motor block and side effects.

ELIGIBILITY:
Inclusion Criteria:

* patients to undergo knee surgery

Exclusion Criteria:

* patients with coagulopathy
* pregnant
* infection at the puncture site
* chronic pain

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Pain Scores on the Visual Analog Scale | two years
  45 patients classified as ASA P1 or P2 aged between 18 and 65 candidates for elective knee operation via arthroscopy were included in the study. All patients received femoral nerve block guided by ultrasound with bupivacaine, 22 ml. The first patient at a concentration of 0.25%. The other patients with higher or lower concentrations if the first patient has pain> 3 or <3 on visual analogic scale respectively after awakening of surgical anesthesia. For surgical anesthesia each patient will undergo general anesthesia. At the end of the surgical procedure and anesthetic awakening patients will be evaluated for analgesia by verbal numeric scale. The modified Dixon method was used to find the EC50 and EC95 of bupivacaine for analgesia of femoral nerve block guided by ultrasound. Concentration still correlated with motor block and side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Ed Carlos Moura, research, Principal Investigator — Federal University of São Paulo
Locations (1):
- Universidade Federal de São Paulo, São Paulo, São Paulo, Brazil